CLINICAL TRIAL: NCT05723237
Title: The Effect of Breast Cancer Screening Training Given to Municipal Women on Health Literacy, Breast Cancer Screening Beliefs and Behaviors
Brief Title: The Effect of Breast Cancer Screening Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, DİLEK YILDIRIM, Principal Investigator, Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Health Literacy of Breast Ca
Record Dates: First submitted 2023-02-03; First posted 2023-02-10 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Women's Health: Neoplasm of Breast

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): The women in the experimental group (n=60) will be given 16 hours of breast cancer screening training, two days a week, two hours a day (60 min+60 min) for four weeks, by the researchers.
  Interventions: Other: Breast Cancer Education
- Control Group (No Intervention): No application will be made to the control group (n=60).

INTERVENTIONS:
Other: Breast Cancer Education — The women in the experimental group (n=60) will be given 16 hours of breast cancer screening training, two days a week, two hours a day (60 min+60 min) for four weeks, by the researchers.
  Arms: Experiment

SUMMARY:
The lack of knowledge of women on breast cancer and health literacy poses a major obstacle to people's breast cancer screening behaviors and beliefs. In order to increase social sensitivity and awareness on this issue; In particular, it is important to research, examine and examine how the municipalities and their employees, who are representatives of the society, evaluate breast cancer screening studies. The aim of our project is to evaluate the effect of breast cancer screening training given to women working in the municipality on health literacy, breast cancer screening belief and behavior. This study will be conducted in a randomized-controlled experimental design with women (n=120) working in a municipality in Istanbul Province between November 2022 and November 2023. Data will be obtained face-to-face using the Participant Information Form, the Health Literacy Scale and the Breast Cancer Screening Beliefs Scale. The women in the experimental group (n=60) will be given 16 hours of breast cancer screening training, two days a week, two hours a day (60 min+60 min) for four weeks, by the researchers. No application will be made to the control group (n=60). Follow-up evaluations of the research will be completed in the following six months. The Health Literacy Scale and Breast Cancer Screening Beliefs Scale will be re-administered to all women in the experimental and control groups at the first follow-up after three months and at the second follow-up after 6 months. The data will be analyzed with statistical methods and the effectiveness of the training will be evaluated.

When the project is concluded; The results will be presented as an article in a national or international journal, or as an oral presentation at a national or international congress. It will be ensured that breast cancer screening training given to women working in the municipality will increase their level of health literacy, have a positive effect on breast cancer screening belief and behavior, and increase their awareness and knowledge level on this subject. In the long term, widespread effects such as reducing the costs women spend on breast cancer, reducing mortality and morbidity rates, raising a conscious society, training undergraduate students involved in the project, and helping them learn by experiencing the research conducted at the national level are foreseen.

DETAILED DESCRIPTION:
Breast cancer is a disease that occurs with the uncontrolled proliferation of cells surrounding the milk glands and ducts in the breast. According to the 2020 data of the International Agency for Research on Cancer (IARC) Global Cancer Obsevartory (GLOBOCAN); The most common type of cancer among women worldwide is breast cancer. At the same time, breast cancer ranks second among deaths of known cause (IARCH, 2020). Similarly, according to 2019 data from the Health Statistics Yearbook, breast cancer ranks first among the most common cancer types among women in Turkey, and ranks second among deaths of known cause.

Early diagnosis in breast cancer is of great importance in increasing the survival rate and increasing the success of treatment. The fact that risk factors are effective in 20% of breast cancer cases and that most of these factors are unchangeable risk factors increases the importance of early diagnosis. Thanks to breast cancer screening methods, it is the first priority to catch breast cancer at an early stage before the clinical signs of breast cancer manifest itself and to reduce mortality rates. Early detection screenings such as Breast Self Examination (BSE), Clinical Breast Examination (CBE), and mammography are thought to be a way to increase early detection and decrease mortality rates.. According to the Turkish National Breast Cancer screening criteria, women older than 20 should periodically perform BSE every month; It is stated that women in the 20-40 age group should have CBE once every two years and women in the 40-69 age group should have CBE once a year. It is also recommended that all women between the ages of 40-69 have a mammogram every two years.

In detecting cancer at an early stage, it is extremely important to have information about the symptoms of cancer and to transform this information into behavior and observe in terms of symptoms. It is suggested that preventive behaviors such as a healthy lifestyle and health screening are beneficial methods in the prevention of breast cancer. In the literature, it has been determined that the knowledge level of women about cancer is not sufficient and they do not participate in breast cancer screening programs at the desired level and periodically.

Studies have also reported that women's attitudes towards breast cancer prevention behaviors and their level of knowledge are related to health literacy. Health literacy is extremely important for the health and health services of the general population because of its consequences that affect individuals and public health. Health literacy level, which is one of the factors that shape women's health, is effective in improving and managing women's health, and understanding and using the necessary information about women's health also increases the behavior of providing early diagnosis against diseases.. A high level of health literacy plays an important role in the protection of public health, as it constitutes an integral part of preventive health services as well as increasing the quality of life and eliminating inequalities. Considering the results of a study conducted in our country; It has been found that 68.9% of the individuals forming the society have insufficient or problematic-limited, 23.4% sufficient and 7.7% excellent health literacy level. Since individuals with low health literacy levels have difficulty in making the right decision about their health, their attitudes and behaviors towards cancer screening are more inadequate. In a study conducted in Turkey, it was concluded that women with limited health literacy had a low level of breast cancer knowledge, and that the low level of economic status and education also affected this situation. For this reason, low health literacy is considered as an important issue in terms of improving individuals' breast cancer knowledge levels and attitudes and behaviors towards screening. In a study, it was concluded that not performing BSE and not having mammography were associated with low health literacy levels. In another study, it is reported that the rate of women not having a mammogram is 52.2% and those who do not have a mammogram have a lower level of health literacy compared to women who have had a mammogram at least once.

As can be seen from the results of the study, the lack of knowledge of women on breast cancer and health literacy poses a major obstacle to people's breast cancer screening behaviors and beliefs. In order to increase social sensitivity and awareness on this issue; In particular, it is important to research, examine and examine how the municipalities and their employees, who are representatives of the society, evaluate breast cancer screening studies. From this point of view, we aimed to evaluate the effect of breast cancer screening training given to women working in the municipality on health literacy, breast cancer screening belief and behavior in our project.

With this training, awareness of women working in the municipality about breast cancer will be raised and it will be contributed to the municipalities, which are representatives of the society, to take steps to make programs that can reach a wider population. In addition, it is thought that this study will contribute to studies evaluating the effect of breast cancer screening education, which is limited in the literature, on health literacy, breast cancer screening belief and behavior.

Breast cancer is the second most common cause of death in our country and in the world. Early diagnosis in breast cancer is of great importance in increasing the survival rate and increasing the success of treatment. Studies have shown that women's knowledge about cancer is not at a sufficient level, they do not participate in breast cancer screening programs at the desired level and periodically, and their health literacy level is insufficient. The reason for this inadequacy is the lack of information. Many educational programs on breast cancer are organized. However, these programs are usually daily or weekly and are limited to increasing the level of knowledge. Breast cancer screening training cannot turn into behavior. With this study, the participants will be monitored for at least 6 months, and an effective fight against breast cancer will be taken. With the study, the knowledge and awareness of the employees working in municipalities, which are representative of the society, will be created through training and education on breast cancer screening. The results of our study will contribute to public health and to reduce health costs by preventing breast cancer with early diagnosis, with the increase in breast cancer screening rates in the long term. Nurses who play a leading role in public health and we, nurse candidates, will contribute to take steps in making programs that can reach a wider population in this regard.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 and over,
* Volunteering to participate in the study,
* Working in the municipality for at least 1 month and
* Not having any communication problems

Exclusion Criteria:

* Women who have any communication barrier and
* Do not volunteer to participate in the study will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Information Form | 1. day
  It includes demographic information such as age, education level, income level, occupation, and duration of employment. In addition, it includes questions about whether they have sufficient information about breast cancer screening, whether they have received education, smoking status, and whether they have a chronic disease.
Health Literacy Scale | 1. day
  It is a five-point Likert scale containing 25 items. There is a positive relationship between the total score obtained from the scale and health literacy, and as the score obtained from the scale increases, the health literacy level of individuals also increases. It consists of four sub-dimensions. The first sub-dimension, Access to Information, consists of five items (1-5). The Comprehension of Information sub-dimension consists of seven items (items 6-12). The Evaluation/Evaluation sub-dimension consists of eight items (items 13 to 20). The Application/Using sub-dimension includes five items (items 21-25). The minimum score that can be obtained from the scale is 25; The maximum is 125 points.
Health Literacy Scale | 30th day
  It is a five-point Likert scale containing 25 items. There is a positive relationship between the total score obtained from the scale and health literacy, and as the score obtained from the scale increases, the health literacy level of individuals also increases. It consists of four sub-dimensions. The first sub-dimension, Access to Information, consists of five items (1-5). The Comprehension of Information sub-dimension consists of seven items (items 6-12). The Evaluation/Evaluation sub-dimension consists of eight items (items 13 to 20). The Application/Using sub-dimension includes five items (items 21-25). The minimum score that can be obtained from the scale is 25; The maximum is 125 points.
Health Literacy Scale | 60th day
  It is a five-point Likert scale containing 25 items. There is a positive relationship between the total score obtained from the scale and health literacy, and as the score obtained from the scale increases, the health literacy level of individuals also increases. It consists of four sub-dimensions. The first sub-dimension, Access to Information, consists of five items (1-5). The Comprehension of Information sub-dimension consists of seven items (items 6-12). The Evaluation/Evaluation sub-dimension consists of eight items (items 13 to 20). The Application/Using sub-dimension includes five items (items 21-25). The minimum score that can be obtained from the scale is 25; The maximum is 125 points.
Breast Cancer Screening Beliefs Scale | 1. day
  The scale consists of 13 items. The scale consists of three sub-dimensions. Attitude towards health screenings sub-dimension items 1, 2, 3 and 4, breast cancer knowledge and perceptions sub-dimension items 5, 6, 7 and 8, and obstacles for mammography screenings sub-dimension 9, 10, 11, 12 and 13 consists of substances.The lowest score obtained from the scale is 0, and the highest score is 100. The fact that the mean score of the sub-dimensions of the scale is 65 and above indicates that screening beliefs have increased positively, their level of knowledge has increased and the barriers to mammography screening have decreased.
Breast Cancer Screening Beliefs Scale | 30th day
  The scale consists of 13 items. The scale consists of three sub-dimensions. Attitude towards health screenings sub-dimension items 1, 2, 3 and 4, breast cancer knowledge and perceptions sub-dimension items 5, 6, 7 and 8, and obstacles for mammography screenings sub-dimension 9, 10, 11, 12 and 13 consists of substances.The lowest score obtained from the scale is 0, and the highest score is 100. The fact that the mean score of the sub-dimensions of the scale is 65 and above indicates that screening beliefs have increased positively, their level of knowledge has increased and the barriers to mammography screening have decreased.
Breast Cancer Screening Beliefs Scale | 60th day
  The scale consists of 13 items. The scale consists of three sub-dimensions. Attitude towards health screenings sub-dimension items 1, 2, 3 and 4, breast cancer knowledge and perceptions sub-dimension items 5, 6, 7 and 8, and obstacles for mammography screenings sub-dimension 9, 10, 11, 12 and 13 consists of substances.The lowest score obtained from the scale is 0, and the highest score is 100. The fact that the mean score of the sub-dimensions of the scale is 65 and above indicates that screening beliefs have increased positively, their level of knowledge has increased and the barriers to mammography screening have decreased.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydin University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No